CLINICAL TRIAL: NCT06712147
Title: A Promotora-centric Community Collaborative to Improve Connections to Mental Health Service
Brief Title: MHE3 Clinical Trial - Overcoming Obstacles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jennifer A. Newberry, Associate Professor of Emergency Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 77672; 5R01MD018201-03 (NIH)
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Services; Community Mental Health Services; Community Health Services; Preventive Health Services; Counseling; Community Networks; Community Participation; Hispanic or Latino
Keywords: mental health; promotores de salud; help-seeking; community resources
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental health use, education, and skill-building (Experimental): Participants randomly assigned to this arm will attend a 6 week educational series that will cover topics around mental health.
  Data will be collected form participants at baseline (before the start of the first session), 1 week after the last session, and at 3- and 6- months after the sessions (follow ups).
  Interventions: Behavioral: Overcoming Life's Hurdles: Mental health education
- Resources in the community (Active Comparator): Participants randomly assigned to this arm will attend a 6 week educational series that will cover topics on resources in the community.
  Data will be collected form participants at baseline (before the start of the first session), 1 week after the last session, and at 3- and 6- months after the sessions (follow ups).
  Interventions: Behavioral: Overcoming Life's Hurdles: Resources in the community

INTERVENTIONS:
Behavioral: Overcoming Life's Hurdles: Mental health education — The intervention group will cover educational topics around mental health including: mental health literacy, individual coping skills, stigma reduction strategies, resources for mental health support, and mental health rights.
  Arms: Mental health use, education, and skill-building
Behavioral: Overcoming Life's Hurdles: Resources in the community — The control group will cover topics including: mental health resources in the community, violence (i.e. domestic violence), employment and education opportunities, housing and tenant rights, immigration and acculturation, and community team building and empowerment.
  Arms: Resources in the community

SUMMARY:
The goal of this clinical trial is to increase and strengthen connections between Latinx individuals and mental health services. Through this intervention, the investigators aim to improve mental health literacy, decrease stigma, increase coping skills, and increase mental health help seeking, even before they are in crisis. Participants will be asked to participate in six educational sessions hosted by Promotores de Salud.

ELIGIBILITY:
Inclusion criteria:

* Has heritage or self-identifies as Hispanic, Latino/a, or Latinx/e
* Must speak English or Spanish
* Primary residence is in 95116, 95122, 95127, 95112, 95111, 95121,95148, or 95133 zip codes

Exclusion criteria:

* Persons from the same household
* First degree family member

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Attitudes Toward Seeking Professional Psychological Help Scale - Short Form | 6 month follow up
  The ATSPPH-SF is scored 0 to 30. Items are rated on a Likert scale (e.g., strongly disagree to strongly agree), with higher scores indicating greater openness to seeking psychological help.

SECONDARY OUTCOMES:
Mental Health Service Use | 3 month follow up and 6 month follow up.
  Measured through a study-specific, 9-item questionnaire. Self-rated mental health status question will use a multiple choice semantic differential scale ("excellent" to "poor"). Number of poor mental health days in the past month will use a numerical scale (0 to 30 days). Mental health help-seeking questions related to wanting, tried, and successfully seeing a mental health professional will use select all that apply time point response options ("never", "in the past 3 months", "within the last 4- 6 months", "over a year ago").
Attitudes Toward Seeking Professional Psychological Help Scale - Short Form | 1 week follow up and 3 month follow up.
  The ATSPPH-SF is scored 0 to 30. Items are rated on a Likert scale (e.g., strongly disagree to strongly agree), with higher scores indicating greater openness to seeking psychological help.
General Self-Efficacy Scale | 1 week follow up, 3 month follow up, and 6-month follow up.
  Measured through a 10-item questionnaire; assesses the strength of an individuals belief of their ability to respond to novel or difficult situations to deal with any associated obstacles or setbacks. Items are rated on a 4-point Likert scale (e.g., 1 = Not at all true to 4 = Exactly true), with higher scores indicating stronger self-efficacy.
Treatment Expectation Questionnaire | 1 week follow up, 3 month follow up, and 6-month follow up.
  Measured through a 6 item questionnaire; measure's a participants expectations about the effectiveness of their treatment. Items are rated on a Likert scale (e.g., from "not at all" to "very much"), and higher scores indicate stronger positive expectations about the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Newberry, MD, JD, MSc, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through presentations at national scientific meetings, publishing in peer reviewed journals, and uploading the processed data to publicly accessible servers, as appropriate. The investigators will conform with the HIPAA Privacy Rule under which protected health information may be used or disclosed by covered entities for research purposes and protect against the involuntary release of data that could identify research participants as stated in the confidentiality statement.
  In accordance with guidelines set by NIH's Policy for Data Management and Sharing, data from this study will be made publicly available through Stanford's Digital Repository (SDR) and the Center for Open Science's OSF repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code